CLINICAL TRIAL: NCT05084300
Title: Effectiveness Pain Neuroscience Education Program in the Executive Functions and Pain Intensity in Patients With Fibromyalgia.
Brief Title: Effectiveness Pain Neuroscience Education In The Executive Functions In Patients With Fibromyalgia
Acronym: PNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Neurociencia Del Dolor (Other)
Collaborators: Universidad de la Costa, Barranquilla, Colombia (Unknown); Instituto Transdisciplinario de Rehabilitación (ITR), Puebla, México (Unknown); Centro Mexicano Universitario de Ciencias y Humanidades (CMUCH), Puebla, México (Unknown); Centro de Artritis y Osteoporosis, Barranquilla, Colombia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INeurocienciaDolor0001
Record Dates: First submitted 2021-03-18; First posted 2021-10-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia; Executive Function; Neuroscience
Keywords: Pain; Neurophysiology; Education
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (Experimental): Pain neuroscience education in addition medical treatment. Pain neuroscience education can be defined as an educational session or sessions describing the neurobiology and neurophysiology of pain, and pain processing by the nervous system.
  Interventions: Other: Pain Neuroscience Education; Other: Usual care
- Usual care (Other): The control group is treated with usual medication for fibromyalgia, anxiolytics, antidepressants, analgesics, ... Depending on the medical needs and criteria of patients´s primary care physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pain Neuroscience Education — A total of 10 PNE sessions (Neuroscience pain education) will be carried out, two each week in addition medical treatment similar to control group (Usual care). The NPE sessions will be conducted by an experienced NPE certified physical therapist in 35 minute face-to-face group sessions. In NPE, the patient is taught about the physiology of pain, central sensitization, representation of the different body regions in the brain, pain-related changes in body perception, and the psychosocial dimensions of pain.
  Other Names: Pain Neurophysiology Education
  Arms: Pain Neuroscience Education
Other: Usual care — The control group (Usual care) is treated with usual treatment, managment or medication for fibromyalgia, anxiolytics, antidepressants, analgesics. Depending on the medical needs and criteria of patients´s primary care physician.

SUMMARY:
Fibromyalgia (FM) is a chronic, complex and disabling clinical entity that has an average global prevalence of 2.7%. It occurs mainly in women in a 3: 1 ratio. It is characterized by persistent generalized pain, fatigue, unrefreshing sleep, cognitive dysfunction and numerous systemic symptoms such as dizziness, migraine, digestive alterations or sensory intolerances. At present there is no pharmacological treatment with specific indication for FM. Usually, non-curative treatments are recommended that alleviate the symptoms of the patients and improve their quality of life and functionality.

Many studies have shown cognitive impairment in FM patients compared to control groups, and FM patients mainly show problems with working memory processes and / or in their attentional and executive domains, as well as in speed of speech. processing (BD Dick, Verrier, Harker, & Rashiq, 2008; Glass, 2009; Tesio et al., 2015; Williams, Clauw, & Glass, 2011).

Many patients with FM have little understanding of their condition, leading to maladaptive pain cognitions and coping strategies. Current research has suggested the use of physiotherapy and rehabilitation in addition to cognitive patient education in the treatment of fibromyalgia. This study aimed to explore the effectiveness of pain neuroscience education in patients with FM.

Therefore, this research aims to analyze the effectiveness of the neuroscience education program on pain in executive functions and the intensity of pain in patients with FM.

DETAILED DESCRIPTION:
The design of the present study will be a parallel-group randomized controlled trial that will be performed between september 2021 and march 2022.

Total = 62 patients. Experimental: PNE (31), Control: Usal care (31). Experimental: In individualized sessions to 31 patients, a health professional will explain the neurological mechanisms that are behind the perception of pain, fatigue and illness from the recent knowledge in neuroscience about brain and pain, as well as the brain's ability to change patien´s behaviour thanks to neuroplasticity.

There will be 10 sessions of 35 minutes, 2 times per week.

Each week the contents of the class and other complementary materials will be sent to the patients.

He outcomes will be assessed at baseline (t1) and one week after intervention (t2). Written informed consent will be acquired for all participants prior to their participation. The study will be implemented and reported in line with the CONSORT statement.

ELIGIBILITY:
Inclusion Criteria:

* (1) Be female
* (2) Age between 40-60 years.
* (3) Sign the consent form.
* (4) Diagnosis of fibromyalgia, according to the American College of Rheumatology criteria;
* (5) Mini Mental State Examination Score greater than or equal to 26 points
* (6) Schooling of at least 12 years (basic primary and secondary).
* (7) Have Spanish as their native language
* (8) Internet access

Exclusion Criteria:

* (1) Pregnant woman
* (2) Illiterate
* (3) Inflammatory rheumatic disease
* (4) Major neurological or psychiatric disease, Intellectual disability (mental retardation) or learning disorders at the premorbid level or severe language comprehension problems.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale-Pain (EVA) | at baseline and through intervention's completion, 5 weeks.
  The severity of the pain at rest was assessed on a 10 cm visual analog scale (Total score: 0-10)(0=no pain, 10=severe pain) Higher scores mean a worse outcome.
Change in Wisconsin card sorting test (WCST) | at baseline and through intervention's completion, 5 weeks.
  The WCST measures cognitive processes such as administrative control, characterization, perseveration, executive function, conceptualization, abstract thinking and reasoning, and it is mainly linked to frontal lobe .
  Commonly used neuropsychological computerized test to assess the ability to form abstract concepts, to shift and maintain set, and to utilize feedback. Total number of categories completed and perseverative errors (reported as t-score with range <20 to >80) will be reported. Higher values indicate better outcome.
Change in Simon task | at baseline and through intervention's completion, 5 weeks.
  A cognitive task, assessing control processes under speeded conditions, measured by response time and accuracy rate. shorter response time and higher accuracy rate indicate better performance.
Change in Visual-spatial working memory span measured by Corsi Block-Tapping task | at baseline and through intervention's completion, 5 weeks.
  The paradigm was computer-adaptive, and thus the set size would only increase if the participant passed consecutive two trials of the same span. The lowest span level started from 2 (2 squares that change color) and up to 9 as maximum.

SECONDARY OUTCOMES:
Change in Stroop Color-word Task | at baseline and through intervention's completion, 5 weeks.
  In the Stroop, the participant is required to name the color of the ink in which a word is printed while inhibiting the overlearned response of reading the word (e.g., the word ''red'' might be printed in blue ink). The number of errors were subtracted from the time required (RT; Reaction Time) for each of the 3 trials, yielding three summary scores. The derived interference score is obtained by subtracting the RT for the first trial from the RT for the third trial.
Change in Central Sensitization Inventory Score (CSI) | at baseline and through intervention's completion, 5 weeks.
  Central Sensitization Inventory (CSI) is a scale used to detect patients with symptoms associated with central sensitization or types of central sensitization syndrome such as fibromyalgia, temporomandibular joint disease, tension type headache, migraine.
  The Central Sensitization Inventory (CSI) consists of two parts:
  Part A consists of 25 questions about central sensitization syndrome (CNS) symptoms; Section B examines the patient's condition of being diagnosed with certain CNS diseases or CNS related diseases such as anxiety and depression.
  The patient answers 25 questions in section A with a score between 0 and 4. The total score will be between 0-100. Results above 40 points indicate central sensitization.
Change in Pain Catastrophizing Scale (PCS) | at baseline and through intervention's completion, 5 weeks.
  The PCS is measured with a self-administered questionnaire. The Pain Catastrophizing Scale is a 13-item inventory that measures 3 elements of the perception of the intensity of pain (rumination, magnification, feeling helpless). Participants indicate the degree to which they agree with statements related their pain by selecting 0 = not at all, 1 = to a slight degree, 2 = to a moderate degree, 3 = to a great degree, 4 = all the time. There are three subscale scores assessing rumination, magnification and helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel.
Change in Tampa Scale for Kinesiophobia (TSK-11) | at baseline and through intervention's completion, 5 weeks.
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Change in Beck Depression Inventory Score | at baseline and through intervention's completion, 5 weeks.
  Beck Depression Criterion (BDI) is a commonly used evaluation criterion for diagnosis and follow-up parameters in assessing depression status.
  It contains 21 categories to measure physical, emotional, cognitive and motivational symptoms such as hopelessness, irritability, guilt, feeling of punishment, fatigue, and weight loss in each depression, and each category is scored between 0-3. The patient is asked to mark the most appropriate one for the four options in each category. Scoring progressively increases from the absence of symptoms to severe symptoms. 0-10 points: No depression, 11-17 points: Mild depression, 18-23 points: Moderate depression, 24 and above points: Severe depression.

OTHER OUTCOMES:
Change in Fibromyalgia Impact Questionnaire (FIQ) | at baseline and through intervention's completion, 5 weeks.
  The FIQ is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes. A validated self-reported questionnaire developed for FM (scores range from 0 to 100, average FM patients score about 50 and severely affected patients score >70) wich measures multidimensional function/health-related quality of life.
Minimental State Examination Folstein | at baseline and through intervention's completion, 5 weeks.
  Mini-Cognitive Lobo est (MEC). To assess the cognitive status before inclusion in the study, the spanish version of Folstein's Minimental State Examination is used. Adapted and validated by Lobo in Spain in 1979. It is a brief cognitive test that consists of the evaluation of the most important cognitive areas (orientation, concentration, calculation, memory, language and construction) with a global maximum score of 35 (30-35 = normal, 24-29 = borderline, <24 in people over 65). The MEC has widely shown its reliability, validity and discriminative power, with a specificity of 75.1% and a sensitivity of 89.8%.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Lopez, PhD, Study Director — Doctorado en Neurociencia Cognitiva Aplicada, Universidad de la Costa
Locations (2):
- Centro de Artritis y Osteoporosis, Barranquilla, Atlántico, Colombia
- Instituto Transdisciplinario de Rehabilitación (ITR), Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morales-Osorio MA, Ramirez-Velez R, Mejia-Mejia J, Martinez-Martinez LA, Roman F, Lopez-Perez PJ, Ordonez-Mora LT. Efficacy of a pain neuroscience educational program in improving executive function and pain intensity in fibromyalgia patients (Fibrobrain project): Study protocol for a randomized controlled clinical trial. Contemp Clin Trials. 2024 Dec;147:107731. doi: 10.1016/j.cct.2024.107731. Epub 2024 Oct 31. PMID 39486209